CLINICAL TRIAL: NCT03328195
Title: A Pilot Study Evaluating the Feasibility, Safety, and Efficacy of the Vielight Neuro RX Gamma Device for the Treatment of Moderate-to-severe Alzheimer's Disease
Brief Title: Vielight Neuro RX Gamma - Feasibility Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vielight Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P17.02
Record Dates: First submitted 2017-10-06; First posted 2017-11-01 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Neuro RX Gamma synchronous (Active Comparator): Neuro RX Gamma device delivering near infra-red light through four diodes positioned over the scalp and one positioned inside the nostril.The synchronous device delivers a synchronized pulse frequency of 40 Hz from all LED clusters.
  Interventions: Device: Neuro RX Gamma synchronous
- Sham light therapy (Sham Comparator): Sham Neuro RX Gamma device having the same appearance and sound as the Neuro RX Gamma device but does not emit the near-infrared light.
  Interventions: Device: Sham
- Neuro RX Gamma asynchronous (Active Comparator): Neuro RX Gamma device delivering near infra-red light through four diodes positioned over the scalp and one positioned inside the nostril. The asynchronous device alternatively delivers pulses from the intranasal and anterior LEDs vs. from the posterior LEDS.
  Interventions: Device: Neuro RX Gamma asynchronous

INTERVENTIONS:
Device: Neuro RX Gamma synchronous — Twenty minute treatment, six days per week for 12 weeks
  Arms: Neuro RX Gamma synchronous
Device: Sham — Twenty minutes, six days per week for 12 weeks with sham device
  Arms: Sham light therapy
Device: Neuro RX Gamma asynchronous — Twenty minutes, six days per week for 12 weeks with sham device
  Arms: Neuro RX Gamma asynchronous

SUMMARY:
This study tests the effects of the Neuro RX Gamma synchronous and asynchronous devices on the cognitive and behavioral functioning of subjects with moderate-to-severe Alzheimer's Disease. The Neuro RX Gamma is non-invasive and delivers near-infrared energy to the brain in daily treatment sessions at home. An optional substudy will involve the use of the Electroencephalogram (EEG) to assess the effect of the treatment devices on the electrical activity of the brain compared to sham.

DETAILED DESCRIPTION:
The Neuro RX Gamma system is a headset which emits pulsed near-infrared energy synchronously or asynchronously through diodes placed on the scalp and inside a nostril.

A potential participant will undergo screening procedures to confirm eligibility to participate in the study, followed by randomization procedure to one of the study groups - treatment synchronized, treatment asynchronized or sham (placebo). A dedicated caregiver will apply the device to the subject for 20 minute daily sessions at home, 6 days a week for a total of 12 weeks. The subject and caregiver will be required to return to the clinic for follow-up assessments after 3, 6 and 12 weeks of treatment. Participants will have the choice of opting into a substudy involving the collection of rest EEG recordings during the baseline and weeks 3, 6 and 12 visits.

60 patients will be enrolled in 2 clinical sites in Ontario, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Age is greater than or equal to 50 years old
* Meets the criteria for probable Alzheimer's disease of the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA)
* If receiving ongoing cholinesterase inhibitor therapy and/or memantine, must be on a stable dosage for at least the prior 3 months
* Mini Mental State Examination (MMSE) score between 0-20 at screening assessment
* Severe Impairment Battery score at baseline of ≤90
* Outpatient with a reliable caregiver willing to commit to study visits and procedures

Exclusion Criteria:

* Current psychiatric or other neurologic disease
* Any history of stroke, seizures, light sensitivity (polymorphous light eruption, solar urticaria, persistent light reactivity) or Lyme disease, including those taking photosensitizing medication
* Currently undergoing light therapy treatment
* Increased skin sensitivity at the treatment site including active herpes simplex in the treatment area, history of keloid formation, or history of retinoid use in the past month
* Pregnant or lactating or planning to become pregnant
* Any issues with ambulation, vision, or hearing which could, in the opinion of the investigator, interfere with their ability to complete assessments
* Does not speak English at a level necessary for the completion of the assessments.
* Currently participating in another clinical research study involving an investigational product.
* Has participated in a drug or device study within the last 30 days.
* Any condition, such as agitation/aggression, that in the opinion of the investigator would cause the patient to be unable to comply with study procedures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Change in the Severe Impairment Battery (SIB) score - An assessment of Severe Dementia in the elderly. | Baseline to Week 12
  The SIB evaluates cognitive abilities in severely impaired individuals. This scale covers social interaction, memory, orientation, language, attention, praxis, visuospatial ability, construction and orientation to name. There are 40 items and the SIB score ranges from 0-100. Individuals who score less than 63 on the SIB are rated as very severely impaired.

SECONDARY OUTCOMES:
Device safety according to the number of device-related adverse events | Baseline to Week 12
  Subjects will be monitored for clinical evidence of device-related adverse events throughout the study.
Change in the Severe Impairment Battery score - An assessment of Severe Dementia in the elderly. | Baseline to Week 3
  The SIB evaluates cognitive abilities in severely impaired individuals. This scale covers social interaction, memory, orientation, language, attention, praxis, visuospatial ability, construction and orientation to name. There are 40 items and the SIB score ranges from 0-100. Individuals who score less than 63 on the SIB are rated as very severely impaired.
Change in the Severe Impairment Battery score - An assessment of Severe Dementia in the elderly. | Baseline to Week 6
  The SIB evaluates cognitive abilities in severely impaired individuals. This scale covers social interaction, memory, orientation, language, attention, praxis, visuospatial ability, construction and orientation to name. There are 40 items and the SIB score ranges from 0-100. Individuals who score less than 63 on the SIB are rated as very severely impaired.
Change in the Alzheimer's Disease Cooperative Study - Activities of Daily Living for Severe Alzheimer's Disease (ADL SAD) score | Baseline to Week 3
  The ADL SAD assesses the performance of activities of daily living by patients with Alzheimer's disease. The assessment includes 19 questions. The score for each question ranges as follows: questions 1 - 5, 0 - 15; questions 6 - 8, 0 - 13; questions 9 - 12, 0 - 12; questions 13 - 15, 0 - 10 and questions 16 - 19, 0 - 4. Subscales will be summed to compute the total score. The total score ranges from 0 - 54 with higher scores indicating less functional impairment and greater competence.
Change in the Alzheimer's Disease Cooperative Study - Activities of Daily Living for Severe Alzheimer's Disease (ADL SAD) score | Baseline to Week 6
  The ADL SAD assesses the performance of activities of daily living by patients with Alzheimer's disease. The assessment includes 19 questions. The score for each question ranges as follows: questions 1 - 5, 0 - 15; questions 6 - 8, 0 - 13; questions 9 - 12, 0 - 12; questions 13 - 15, 0 - 10 and questions 16 - 19, 0 - 4. Subscales will be summed to compute the total score. The total score ranges from 0 - 54 with higher scores indicating less functional impairment and greater competence.
Change in the Alzheimer's Disease Cooperative Study - Activities of Daily Living for Severe Alzheimer's Disease (ADL SAD) score | Baseline to Week 12
  The ADL SAD assesses the performance of activities of daily living by patients with Alzheimer's disease. The assessment includes 19 questions. The score for each question ranges as follows: questions 1 - 5, 0 - 15; questions 6 - 8, 0 - 13; questions 9 - 12, 0 - 12; questions 13 - 15, 0 - 10 and questions 16 - 19, 0 - 4. Subscales will be summed to compute the total score. The total score ranges from 0 - 54 with higher scores indicating less functional impairment and greater competence.
Change in the Neuropsychiatric Inventory (NPI) score which assesses behavioral changes in neurologic illnesses based on a standardized caregiver interview. | Baseline to Week 3
  The NPI assesses the frequency, severity and level of distress caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and appetite/eating).
Change in the Neuropsychiatric Inventory (NPI) score which assesses behavioral changes in neurologic illnesses based on a standardized caregiver interview. | Baseline to Week 6
  The NPI assesses the frequency, severity and level of distress caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and appetite/eating).
Change in the Neuropsychiatric Inventory (NPI) score which assesses behavioral changes in neurologic illnesses based on a standardized caregiver interview. | Baseline to Week 12
  The NPI assesses the frequency, severity and level of distress caused by 12 common dementia-related behaviors (delusions, hallucinations, agitation/aggression, depression/dysphoria, anxiety, elation/euphoria, apathy/indifference, disinhibition, irritability/lability, aberrant motor behavior, sleep and appetite/eating).
Change in the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS CGIC) score. | Baseline to Week 3
  The ADCS CGIC gives the Clinician's assessment of the patient's response to the treatment. It is intended to be used as a measure of clinically meaningful change. The ADCS-CGIC focuses on clinicians' observations of change in the patient's cognitive, functional, and behavioral performance since the beginning of a trial. It relies on both direct examination of the patient and interview of the caregiver. Scored as marked/moderate/minimal improvement or worsening or no change.
Change in the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS CGIC) score. | Baseline to Week 6
  The ADCS CGIC gives the Clinician's assessment of the patient's response to the treatment. It is intended to be used as a measure of clinically meaningful change. The ADCS-CGIC focuses on clinicians' observations of change in the patient's cognitive, functional, and behavioral performance since the beginning of a trial. It relies on both direct examination of the patient and interview of the caregiver. Scored as marked/moderate/minimal improvement or worsening or no change.
Change in the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS CGIC) score. | Baseline to Week 12
  The ADCS CGIC gives the Clinician's assessment of the patient's response to the treatment. It is intended to be used as a measure of clinically meaningful change. The ADCS-CGIC focuses on clinicians' observations of change in the patient's cognitive, functional, and behavioral performance since the beginning of a trial. It relies on both direct examination of the patient and interview of the caregiver. Scored as marked/moderate/minimal improvement or worsening or no change.
Change in the Electroencephalogram's (EEG) overall power spectral density | Baseline to Week 12
  The EEG recordings will give insight into the effect on the neural activity of the brain of the Neuro RX Gamma synchronized and Neuro RX Gamma asynchronized compared to sham.

OTHER OUTCOMES:
Caregiver reported treatment compliance | 12 weeks
  Caregivers will document treatment sessions in a logbook to monitor compliance.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Memory Program, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No